CLINICAL TRIAL: NCT07300358
Title: BIOCLOSE-PFO Study：Evaluation of the Safety and Efficacy of a Biodegradable Patent Foramen Ovale Occluder System: A Prospective, Multicenter, Randomized Controlled, Non-Inferiority Clinical Study
Brief Title: Study on the Safety and Effectiveness of a Biodegradable Patent Foramen Ovale Occluder System
Acronym: BIOCLOSE-PFO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Lingsi Medical Technology Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ShanghaiLingsiMedTech
Record Dates: First submitted 2025-09-15; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Cardiovascular Diseases; Cardiovascular Abnormality; Heart Defects, Congenital; Heart Septal Defects; Heart Septal Defects, Atrial; Foramen Ovale, Patent; Stroke, Ischemic; Stroke (CVA) or TIA
MeSH Terms: conditions — Cardiovascular Diseases; Cardiovascular Abnormalities; Heart Defects, Congenital; Heart Septal Defects; Heart Septal Defects, Atrial; Foramen Ovale, Patent; Ischemic Stroke; Stroke

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cardi-o-fix PFO occluder (Active Comparator): Participants treated with th with the Cardi-o-fix PFO occluder according to the INSTRUCTIONS for Use (IFU)
  Interventions: Device: Active Comparator
- Biodegradable PFO occluder system (Experimental): Participants treated with th with the biodegradable PFO occluder system according to the INSTRUCTIONS for Use (IFU)
  Interventions: Device: Experimental

INTERVENTIONS:
Device: Active Comparator — Percutaneously occlusion of PFO with Cardi-o-fix PFO occluder
  Other Names: Cardi-o-fix PFO occluder
  Arms: Cardi-o-fix PFO occluder
Device: Experimental — Transcatheter closure of a patent foramen ovale (PFO) with biodegradable PFO occluder
  Arms: Biodegradable PFO occluder system

SUMMARY:
To evaluate the Safety and Efficacy of a Novel Biodegradable Occluder for Percutaneous Closure of Patent Foramen Ovale (PFO)

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized, controlled, non-inferiority clinical study. The study aims to evaluate the safety and efficacy of a novel biodegradable patent foramen ovale (PFO) occluder system compared to a conventional metallic occluder in patients with a PFO that is clinically determined to be associated with an PFO⁃associated stroke（PFO-AS）or transient ischemic attack (TIA).

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65 years.
* Presence of a patent foramen ovale (PFO) confirmed by transthoracic echocardiography (TTE) or transesophageal echocardiography (TEE).
* Presence of a moderate-to-large right-to-left shunt (RLS) at rest or during the Valsalva maneuver, as confirmed by agitated saline contrast echocardiography (also known as bubble study).
* Clinically diagnosed with a PFO-associated ischemic stroke or transient ischemic attack (TIA).

Exclusion Criteria:

* An alternative, clearly identified cause of ischemic stroke or TIA (other than PFO) is determined by the investigator.
* Large territory cerebral infarction within 4 weeks prior to the planned procedure.
* Atherosclerotic stenosis (>50%) of the carotid or vertebral arteries, as confirmed by CT angiography or vascular ultrasound per investigator assessment.
* Presence of intracardiac thrombus or vegetation as confirmed by echocardiography.
* Left ventricular ejection fraction (LVEF) < 35%.
* Atrial fibrillation or atrial flutter.
* Left ventricular aneurysm or severe regional wall motion abnormality.
* Significant valvular stenosis or regurgitation, or history of valvular replacement or repair surgery.
* Pulmonary hypertension or a PFO constituting a special conduit (e.g., right-to-left shunt due to elevated right heart pressures).
* Other confirmed causes of right-to-left shunt, such as atrial septal defect (ASD) or pulmonary arteriovenous fistula.
* Complex PFO anatomy (e.g., multi-tunnel PFO) or PFO associated with an ASD requiring different closure strategy.
* Thrombus, mass, or vegetation identified at the intended implant site or along the potential delivery pathway.
* Acute myocardial infarction or unstable angina within 3 months prior to the procedure.
* Previous implantation of an inferior vena cava filter, PFO closure device, or ASD closure device.
* Any other condition deemed by the investigator to make the patient unsuitable for PFO device implantation.
* Concomitant cardiac anomalies requiring surgical correction.
* Uncontrolled systemic or local infection, or sepsis.
* Active infection requiring concurrent antibiotic therapy (Patients with transient conditions may be enrolled after completing antibiotic therapy and a subsequent 14-day washout period).
* Contraindication to antiplatelet or anticoagulant therapy (e.g., major bleeding within 3 months, known retinopathy, history of intracranial hemorrhage, or other significant intracranial pathology).
* Known hypersensitivity or allergy to tantalum or nickel.
* Pregnancy, lactation, or women of childbearing potential not using highly effective contraception.
* Life expectancy less than 1 year due to malignancy or other comorbid disease.
* Current participation in another investigational drug or device clinical study that has not yet completed its primary endpoint.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Success rate of effective occlusion | at 12 months post-implantation
  Effective occlusion was defined as: 12 months after the procedure, Echocardiographyshowed that the position and shape of the occluder were normal, and no horizontal atrial shunt was observed. Re-examination by Contrast echocardiography (cTTE or cTEE) showed no or only a small amount of right-to-left shunt, that is, no microvesicles or less than 10 microvesicles/frame in left heart cavity after Valsalva and resting state.

SECONDARY OUTCOMES:
Success rate of effective occlusion | at 6 months post-implantation
  Effective occlusion was defined as: 6 months after the procedure, Echocardiographyshowed that the position and shape of the occluder were normal, and no horizontal atrial shunt was observed. Re-examination by Contrast echocardiography (cTTE or cTEE) showed no or only a small amount of right-to-left shunt, that is, no microvesicles or less than 10 microvesicles/frame in left heart cavity after Valsalva and resting state.
Device Success Rate | immediately after the procedure
  Successful intraoperative deployment of the occluder, with immediate post-procedure echocardiography confirming appropriate device morphology and position, absence of new pericardial effusion or valvular regurgitation, and successful retrieval of the delivery system
Procedural success Rate | at discharge or 7 days post-procedure
  Successful device implantation without any procedure- or device-related complications prior to discharge. Complications include atrial fibrillation, other serious arrhythmic events, thrombosis, cerebral embolism, pericardial effusion, cardiac tamponade, device embolization, or displacement
Recurrence or incidence of cryptogenic stroke or TIA | From attempted procedure up to 12 months post-implantation
  Cryptogenic stroke was defined as a new focal cerebral ischemia confirmed by neuroimaging (cranial MRI or CT), which was performed After extensive vascular, cardiac, and blood evaluation, non-atherosclerotic, cardiogenic, or arteriolar obliterators were identified Cerebral infarction caused by the diagnosis of exclusion.
All-cause mortality | From attempted procedure up to 12 months post-implantation
  All-cause death is defined as death from any cause during the follow-up period
Incidence of new atrial fibrillation and atrial flutter | From attempted procedure up to 12 months post-implantation
  atrial fibrillation and atrial flutter
Incidence of device-related serious adverse events | From attempted procedure up to 12 months post-implantation
  including but not limited to: Device-related thrombosis、embolic stroke、peripheral arterial embolism、Ⅲ° atrioventricular block、cardiac erosion、infective endocarditis、severe hemolytic anemia
Device defects | From attempted procedure up to 12 months post-implantation
  Device defects refer to unreasonable risks that may endanger human health and safety under normal use of medical devices in clinical trials, such as label errors, quality problems and failures.
Migraine Headache events | At 6 months and 12 months post-implantation
  Change in the number of monthly migraine days from baseline to 6 months and 12 months.
  Change in the number of migraine attacks from baseline to 6 months and 12 months.
  Change in the Score of HIT-6 or VAS or MIDAS from baseline to 6 months and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: XiangBin Pan, Doctor, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital

IPD SHARING:
Plan to Share IPD: No